CLINICAL TRIAL: NCT00158223
Title: Pimozide Augmentation of Clozapine in Schizophrenia
Brief Title: Effectiveness of Pimozide in Augmenting the Effects of Clozapine in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joseph Friedman, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 02-0517; R01MH067806 (NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; Clozapine; Treatment; Combination; Unresponsive; Schizoaffective Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Pimozide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Participants will receive encapsulated placebo made to match active drug
  Interventions: Drug: Placebo
- pimozide (Experimental): Participants will receive pimozide flexible dosing
  Interventions: Drug: Pimozide

INTERVENTIONS:
Drug: Pimozide — Each capsule of active treatment will contain 2 mg of pimozide. Dosing will be flexible and will range from a minimum of 2 mg per day to 8 mg per day. Dosing will begin at Week 1 with 1 capsule per day. This will be slowly titrated at a rate of 1 capsule per week to a maximum of 4 capsules depending upon clinical response and side effects.
  Other Names: Orap
  Arms: pimozide
Drug: Placebo — Active drug and placebo will be encapsulated in an identical fashion. The placebo capsule will be made to match in appearance and weight. There will be flexible dosing, allowing a minimum of 1 capsule per day to 4 capsules per day, in order to match the dosing range of the active treatment.
  Other Names: Sugar Pill
  Arms: placebo

SUMMARY:
This study will assess the effectiveness of pimozide in enhancing the effects of clozapine in the treatment of schizophrenia.

DETAILED DESCRIPTION:
A significant number of schizophrenics exhibit partial or no response to typical antipsychotic medications. Clozapine has been shown to be more effective in treating schizophrenia than typical antipsychotic drugs. However, only an estimated 30% to 60% of people who are unresponsive to treatment with typical antipsychotics will respond to treatment with clozapine. Taking clozapine with pimozide, an antipsychotic drug, can increase clozapine's effects. However, sufficient research on this approach has not yet been performed. This study will assess the effectiveness of pimozide in enhancing the effects of clozapine in the treatment of schizophrenia.

Participants in this double-blind study will receive a stable dose of clozapine for eight weeks prior to enrollment. For the first 4 weeks following enrollment, baseline measurements will be taken. Once a week, participants will report to the study site, where symptom severity, cognitive ability, and functional status, including reading level, will be assessed. In addition, participants will receive a standard medical examination, which will include blood tests and an EKG. Upon completion of this initial phase, participants will be randomly assigned to one of two treatment groups: clozapine combined with pimozide; or clozapine combined with placebo. This phase will last for 12 weeks. Study visits will continue to occur weekly, and will be used to re-assess the measurements obtained during baseline. In addition, participants will have an EKG at each study visit for the first 4 weeks of treatment. All baseline measurements will be repeated in Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV criteria
* Any schizoaffective disorder or subtype
* Score greater than 60 on the Positive and Negative Syndrome Scale (PANSS)
* Currently taking clozapine
* Score of four or higher on two or more items from the positive symptom subscale of the PANSS
* Score of 4 or greater on the Clinical Global Impression (CGI) scale
* Clozapine plasma level greater than 378 µg/ml
* Stable dose of clozapine demonstrated to have been associated with a clozapine plasma level greater than 378 µg/ml for at least eight weeks
* Able to read at an 8th grade level or above

Exclusion Criteria:

* History of unstable coronary artery disease
* Congestive heart failure
* History of long Q-T syndrome
* History of cardiac arrhythmia
* History of cardiac conduction delay
* Baseline QT correction score greater than 0.425 seconds
* Liver disease
* History of stroke
* History of Neuroleptic Malignant Syndrome
* Hypokalemia
* Hypocalcemia
* Current blindness, deafness, language difficulties, or any other disability which may prevent participation or cooperation in the study
* Current suicidal or homicidal thoughts
* Currently abusing psychoactive substances
* Currently receiving antidepressants, thymoleptics, L-DOPA, buspirone, or antipsychotics other than clozapine (Valproic acid and Divalproex sodium are not criteria for exclusion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph I. Friedman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Manhattan Psychiatric Center, New York, New York
  - Pilgrim Psychiatric Center, W. Brentwood, New York

REFERENCES:
- [Background] Friedman J, Ault K, Powchik P. Pimozide augmentation for the treatment of schizophrenic patients who are partial responders to clozapine. Biol Psychiatry. 1997 Sep 15;42(6):522-3. doi: 10.1016/S0006-3223(97)00227-8. No abstract available. PMID 9285089
- [Result] Friedman JI, Lindenmayer JP, Alcantara F, Bowler S, Parak M, White L, Iskander A, Parrella M, Adler DN, Tsopelas ND, Tsai WY, Novakovic V, Harvey PD, Davis KL, Kaushik S. Pimozide augmentation of clozapine inpatients with schizophrenia and schizoaffective disorder unresponsive to clozapine monotherapy. Neuropsychopharmacology. 2011 May;36(6):1289-95. doi: 10.1038/npp.2011.14. Epub 2011 Feb 23. PMID 21346734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from inpatient and outpatient treatment settings at Mount Sinai Hospital, Pilgrim Psychiatric Center and Manhattan Psychiatric Center in New York.
Pre-assignment Details: 16 subjects were excluded during the 4-week symptom stability-screening period before randomization because of withdrawal of consent or a failure to meet inclusion and exclusion criteria. Seven additional subjects were randomized to a haloperidol adjunctive pilot study.
Groups:
- Placebo: Participants received encapsulated placebo made to match active drug
- Pimozide: Participants received pimozide flexible dosing
Period: Overall Study
Arm/Group | Placebo | Pimozide
Started | 28 | 25
Completed | 23 | 22
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimozide | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (8.7) | 45.5 (10.2) | 44.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 20 | 21 | 41
Treatment Setting [Number; unit: participants]
  Inpatient | 19 | 15 | 34
  Outpatient | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Positive Syndrome Scale (PANSS) Total Score
Description: Severity of positive schizophrenic symptoms The Positive Syndrome Scale of the PANSS is comprised of seven items measuring positive such symptoms such as hallucinations, delusions, grandiosity, etc. Each item is scored on a 7 point scale of that particular symptom's severity, ranging from 1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate severe, 6 = severe, and 7 = extreme. The PANSS Positive Subscale seven items has a range of a summed score from 7 (absent) to 49 (extreme psychopathology). Therefore, the higher the score, the more severe the symtpoms.
Time Frame: Variable change from baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pimozide
Number analyzed (Participants) | 23 | 22
units on a scale | -1.05 (2.98) | -1.30 (2.56)

2. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: The Clinical Global Impression-improvement (CGI-improvement) scale is a research rating tool, developed for use in NIMH-sponsored clinical trials provides a brief assessment of the clinician's view of the patient's overall clinical improvement prior to and after initiating a study medication. The CGI-change is rated on a seven point scale ranging from 1= very much improved since the initiation of treatment to 7=very much worse since the initiation of treatment. Therefore, a lower score indicates more improvement in symptoms over time.
Time Frame: variable change from baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pimozide
Number analyzed (Participants) | 23 | 22
units on a scale | -0.35 (0.57) | -0.15 (4.97)

3. Primary Outcome: Negative Syndrome Scale (PANSS) Total Score
Description: Severity of negative schizophrenic symptoms, The Negative Syndrome scale is compromised of seven items, each scored on severity with numeric assignments ranging from 1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate severe, 6 = severe, and 7 = extreme. The items which comprise the Negative Syndrome Scale of the PANSS measure things such as emotional withdrawal, apathy, difficulty in abstract thinking, etc. The seven items which comprise the PANSS Negative Subscale has an aggregate range of 7 (absent) to 49 (extreme psychopathology), a higher score indicating more severe symptoms.
Time Frame: Variable change from baseline to week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pimozide
Number analyzed (Participants) | 23 | 22
units on a scale | -1.59 (4.46) | 0.65 (4.65)

ADVERSE EVENTS:
Arm/Group | Placebo | Pimozide
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 5/28 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Pimozide (N=25)
Severe EPS (Nervous system disorders) | 0 (0) | 1 (1)
delirium (Renal and urinary disorders) | 0 (0) | 1 (1)
bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) — exacerbation of hemorrhoidal bleeding
psychotic symptoms (Psychiatric disorders) | 2 (2) | 0 (0)
bigeminy (Cardiac disorders) | 1 (1) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
withdrew consent (Social circumstances) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Neither baseline nor follow-up clozapine plasma concentrations were reported. Possible that one or both groups did not have therapeutic baseline clozapine levels and/or had pharmacokinetic interactions with the study drug changing concentrations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes